CLINICAL TRIAL: NCT05794997
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Propranolol/Carvedilol Versus Atenolol/Bisoprolol/Sotalol
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019P003607-13
Record Dates: First submitted 2023-03-03; First posted 2023-04-03 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Propranolol; Carvedilol; Atenolol; Bisoprolol; Sotalol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propranolol or Carvedilol: Exposure group
  Interventions: Drug: Propranolol or Carvedilol
- Atenolol, Bisoprolol or Sotalol: Reference group
  Interventions: Drug: Atenolol, Bisoprolol or Sotalol

INTERVENTIONS:
Drug: Propranolol or Carvedilol — Propranolol or Carvedilol claim is used as the exposure group.
  Groups: Propranolol or Carvedilol
Drug: Atenolol, Bisoprolol or Sotalol — Atenolol, Bisoprolol or Sotalol claim is used as the reference group.
  Groups: Atenolol, Bisoprolol or Sotalol

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1ltZHHv6AvMkPBbSp_9c0dtQ0XMmBc00d4jaRId5ovaA/edit?usp=sharing or Appendix A (https://drive.google.com/drive/folders/1a-1uRt73kVywEoV8L0cEmDNgaqYEIudT?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2019 (end of data availability).

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. At least 1 inpatient claim or 2 outpatient claims with hypertension diagnosis recorded in 365 days prior to drug initiation

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission in the 365 days prior to the cohort entry date
* 3. Prior use of Propranolol, Carvedilol and Atenolol, Bisoprolol, Sotalol
* 4. Use of Propranolol, Carvedilol and Atenolol, Bisoprolol, Sotalol concomitantly on index date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing Propranolol or Carvedilol to hydrochlorothiazide. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of Propranolol or Carvedilol or Atenolol, Bisoprolol or Sotalol (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 817337 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol or Carvedilol | Atenolol, Bisoprolol or Sotalol
Started | 583870 | 233467
Completed | 222015 | 222015
Not Completed | 361855 | 11452

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol or Carvedilol | Atenolol, Bisoprolol or Sotalol | Total
Number analyzed (Participants) | 222015 | 222015 | 444030
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 222015 | 222015 | 444030
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.77 (6.82) | 74.75 (6.78) | 74.77 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128266 | 127873 | 256139
  Male | 93749 | 94142 | 187891
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 177198 | 176941 | 354139
  Black | 22448 | 22557 | 45005
  Hispanic | 7289 | 7209 | 14498
  Asian | 7954 | 8042 | 15996
  North American Native | 1347 | 1426 | 2773
  Other | 4242 | 4273 | 8515
  Unknown | 1537 | 1567 | 3104
Dementia risk factors [Count of Participants; unit: Participants]
  Anxiety | 32757 | 32295 | 65052
  Bipolar Disorder | 2299 | 2263 | 4562
  Coronary artery disease | 96483 | 96613 | 193096
  Depression | 32918 | 32329 | 65247
  Diabetes | 168274 | 168200 | 336474
  Obesity | 48216 | 48375 | 96591
  Schizophrenia | 1045 | 1064 | 2109

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 298 days (exp), 249 days (ref) 2) 995 days (exp), 981 days (ref) 3) 515 days (exp), 448 days (ref) 4) 307 days (exp), 253 days (ref)
Population: Study cohort after 1:1 propensity score matching
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Propranolol or Carvedilol | Atenolol, Bisoprolol or Sotalol
Number analyzed (Participants) | 222015 | 222015
Incidence rate per 1000 person year
  Analysis 1 | 22.96 [22.48 to 23.45] | 19.84 [19.35 to 20.33]
  Analysis 2 | 26.82 [26.22 to 27.44] | 25.84 [25.25 to 26.45]
  Analysis 3 | 23.03 [22.47 to 23.60] | 20.21 [19.64 to 20.79]
  Analysis 4 | 7.21 [6.95 to 7.49] | 6.47 [6.20 to 6.75]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 298 (for Propranolol and Carvedilol) and 249 (for Atenolol, Bisoprolol, Sotalol)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Propranolol or Carvedilol | Atenolol, Bisoprolol or Sotalol
All-Cause Mortality (participants affected / at risk) | 0/222015 | 0/222015
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/222015 | 0/222015

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05794997/Prot_SAP_000.pdf